CLINICAL TRIAL: NCT02273427
Title: Randomised 3-way Cross-over Phase I Study to Investigate the Effect of Different Food Compositions (Low Fat and High Fat Meal) on Bioavailability of BIIL 284 BS 75 mg Tablet in Healthy Male Volunteers
Brief Title: Effect of Different Food Compositions on Bioavailability of BIIL 284 BS in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 543.5
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — amelubant

ARMS (3):
- BIIL 284 BS fasted (Active Comparator)
  Interventions: Drug: BIIL 284 BS
- BIIL 284 BS with high fat meal (Experimental)
  Interventions: Drug: BIIL 284 BS; Other: high fat meal
- BIIL 284 BS with low fat meal (Experimental)
  Interventions: Drug: BIIL 284 BS; Other: low fat meal

INTERVENTIONS:
Drug: BIIL 284 BS
Other: high fat meal
  Arms: BIIL 284 BS with high fat meal
Other: low fat meal
  Arms: BIIL 284 BS with low fat meal

SUMMARY:
food effect, relative bioavailability, pharmacokinetics, safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy caucasian males as determined by the results of screening, range from 21 to 50 years of age and be within +- 20% of their normal weight (Broca-Index)
* All volunteers will have given their written informed consent in accordance with Good Clinical Practice and local legislation prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial (<= one week prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 ml within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2000-02; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | up to 72 hours after drug administration
Area under the concentration time curve from timepoint zero extrapolated to infinity (AUC-infinity) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Time to Cmax (tmax) | up to 72 hours after drug administration
Area under the concentration time curve from timepoint zero to time of last data point above limit of quantification (AUC-tz) | up to 72 hours after drug administration
Terminal half-life (t1/2) | up to 72 hours after drug administration
Total mean residence time (MRTtot) | up to 72 hours after drug administration
Volume of distribution during terminal phase after oral administration (Vz/F) | up to 72 hours after drug administration
Total clearance after oral administration (CLtot/F) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital functions | up to 8 days after last drug administration
  blood pressure, pulse rate, ECG
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after last drug administration